CLINICAL TRIAL: NCT06085820
Title: The Effect of Birth Ball and Bırth Dance Applied in The First Stage of Labor on Pain, Type of Birth, Maternal Satisfactıon Ond Duration of Labor
Brief Title: The Effect of Birth Ball and Birth Dance Applied in the First Stage of Labor on Some Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ozlemarı003
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pain, Labor; Satisfaction, Patient
Keywords: birth dance; birth ball; childbirth; labor pain; midwife; satisfaction
MeSH Terms: conditions — Labor Pain; Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: There will be three groups in total in the study, one control and two experimental groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (birth ball) (Experimental): Group A
  * Meeting
  * The researcher will introduce himself/herself, provide information about the research and obtain verbal and written consent.
  * Privacy will be ensured
  * After the routine maintenance of the hospital is carried out in the latent phase, the researcher will first introduce the birthing ball to the pregnant women and the movements to be performed will be demonstrated by the researcher.
  Starting from the active phase, movements will be performed for 20 minutes every hour. During the contraction, there will be a break until the contraction ends, and the pregnant woman will be given the opportunity to rest in a comfortable position. The same movements will be applied again. The partograph will be recorded. VAS and VCS will be applied.
  * When the perineum is crowned, the pregnant woman will be taken to the table.
  * SEMSNB will be applied within 1-4 hours after birth.
  Interventions: Behavioral: Experimental (birth ball)
- Experimental (birth dance) (Experimental): Group B
  * Meeting
  * The researcher will introduce himself/herself, provide information about the research and obtain verbal and written consent.
  * Privacy will be ensured
  * The environment will be made suitable
  * The pregnant woman will be asked to wear slippers that make her feel comfortable.
  * Pregnant will be given training on how to perform the birth dance during the latent phase. VCS and VAS will be applied.
  Birth dance practice will be started on the pregnant woman starting from the active phase.
  * Starting from the active phase, the partograph will be recorded.
  * Birth dance cervical dilation will be performed for 20 minutes every hour, in the range of 5-8 cm.
  * At the end of the active phase, VCS and VAS will be applied again. The researcher will be with the pregnant woman throughout the application and labor.
  * When perineum is crowned, the pregnant woman will be taken to the delivery table.
  SEMSNB will be applied within 1-4 hours after birth.
  Interventions: Behavioral: Experimental (birth dance)
- control group (No Intervention): Midwifery Interventions Made to the Control Group
  * The pregnant woman will be greeted politely.
  * The researcher will introduce himself/herself, provide information about the research and obtain verbal and written consent.
  * Privacy will be ensured
  * An introductory information form will be filled out.
  * Routine monitoring and care will be provided by the medical staff working in the delivery room.
  * At the end of each phase (latent, active), GKS and SCS will be applied once.
  * EFM (Electronic Fetal Monitoring) will be applied in each phase.
  * Child Heart Sound (CHS) will be listened to every half hour and recorded on the partograph.
  * Cervical changes will be evaluated with bimanual examination and recorded on the partograph.
  * When the perineum is crowned, the pregnant woman will be taken to the table.
  * NDAMDÖ will be applied to women taken to the postpartum room within a period of 1-4 hours.

INTERVENTIONS:
Behavioral: Experimental (birth ball) — It is a large and firm ball made of soft, thick plastic, inflated with air. It can be easily inflated and deflated, washable, available in different sizes (55-65-75 cm in diameter) and strong enough to carry weight up to 136 kg.
  When the literature was examined, it was seen that birth balls between 55-75cm were generally used in accordance with the intended use. Appropriate ball size will be determined by the participant's height. In order for the pregnant woman to continue balance exercises, she should be allowed to sit on the round birthing ball with her knees and hips at an angle of approximately 90°, with an upright spine.
  birth ball; It is performed in sitting (pelvic rocking movement, forward-backward and right-left rocking, forward-supported sitting, springing movement), kneeling and squatting (hugging the ball and pelvic rocking movement) positions.
  Arms: Experimental (birth ball)
Behavioral: Experimental (birth dance) — Thanks to the birth dance, the expectant mother perceives less pain. In fact, it is known that a change in position is effective in the perception of pain. On the other hand, if the woman focuses on a point other than the pain during the act, it makes it easier for her to perceive the pain less. The low cost of this application increases its usability.
  The most appropriate time for the birth dance is from the active phase of the first phase of labor until the end of this phase . The expectant mother dances with rhythmic movements accompanied by soothing and soothing music with the help of a birth supporter (midwife, relative, spouse or partner). Optionally, sacral massage can be added to the birth dance. In fact, in addition to reducing the pain experienced through freedom of movement, upright position and massage, it is also aimed to provide emotional support to the woman.
  Arms: Experimental (birth dance)

SUMMARY:
Aim: The study was conducted to investigate the effect of birth ball and birth dance practices applied in the first stage of labour on pain, mode of delivery, maternal satisfaction and duration of labour. Material and Method: This study was conducted as a randomised controlled clinical trial between July 2023 and December 2024. The population of the study consisted of pregnant women who applied to Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital Delivery Department between January 2024 and August 2024. The sample group consisted of a total of 104 primiparous pregnant women, 35 A (round ball group), 33 B (birth dance group) and 36 C (control group), who met the inclusion criteria and were determined by power analysis. Data were collected by using 'Descriptive Information Form', 'Verbal Category Scale', 'Visual Analogue Scale', 'Partograph' and 'Maternal Satisfaction in Childbirth Assessment Scale'. Results: In active phase of labour, birth ball and birth dance practice caused a significant decrease in pain perceptions of pregnant women (p<0.05). It was determined that level of cervical dilatation progressed faster in pregnant women who were administered a round birth ball during labour compared to the other groups. It was also determined that application of birth ball and birth dance in labour accelerated level of fetal head descent in the active phase of labour, shortened duration of the active phase, affected the duration and number of contractions and did not affect labour satisfaction according to the cut-off score of the Maternal Satisfaction in Childbirth Assessment Scale.

Conclusion: The application of birth ball and birth dance in the active phase of labour was found to reduce labour pain, accelerate the level of fetal head descent, shorten duration of the active phase, and affect duration and number of contractions.

DETAILED DESCRIPTION:
Birth ball and birth dance practices are among the primary methods used to provide freedom of movement to women during birth. These methods enable the woman to benefit from all the opportunities provided by the upright position and are important in the normal course of action. One of the main points of birth ball and birth dance practices is squatting. Squatting is a posture in which the legs are opened to the sides and the knees are bent. This position facilitates birth by widening the pelvic outlet.

A birthing ball is one of the methods that help mothers cope with labor pain. Exercise with a birthing ball is considered a useful, non-pharmacological strategy The main advantages of birthing ball exercise during pregnancy include postural corrections, relaxation, stretching and strengthening muscles. Sekendiz et al stated that movements performed with a birth ball increase the strength, resistance, flexibility and balance of the trunk, waist and quadriceps muscles. The use of a birth ball and similar non-pharmacological interventions reduce the need for epidural anesthesia, episiotomy and interventional birth. However, no side effects on mother and baby health have been reported

The birthing ball, also known as the Swiss ball and the Petzi ball, was developed in 1963 and has been used in physical applications of neurodevelopmental therapy. Perez and Simkin introduced the birthing ball as a birthing tool to professional birth assistants, midwives, nurses and students who provide childbirth education since the 1980s. Perez (2001) stated that the use of a birth ball during pregnancy and birth is physically beneficial.

Birth dance is one of the non-pharmacological practices that allows freedom of massage and position changes with the support of the spouse/partner. During the birth dance, the pregnant woman puts her hands on her partner's shoulders and performs pelvic tilt movements accompanied by music; His back and sacrum are massaged by his partner.

Dance, one of the non-pharmacological methods used in birth; It may be a way to reduce technological and medical interventions during labor while also promoting the progression of labor. In many cultures, an upright position during labor is common. An upright position and mobility during labor is recommended because this is likely to improve maternal and fetal circulation while also It also increases maternal comfort.

There are studies on birth ball and birth dance in the relevant literature. However, no study comparing birth dance and birth ball applications has been found in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Those who agree to participate in the research, are over 18 years old and speak Turkish,
* Primiparous pregnant women who do not have any physical or chronic disease and are in the latent phase,
* Pregnant women who do not have a risky pregnancy,
* 38-42. gestational age, singleton pregnant women,
* Absence of diagnosed fetal malformations,
* No medical problems at the beginning of the study,
* Amniotic membranes are not opened,
* Women who are at least primary school graduates will be included in the research.

Exclusion Criteria:

* Pregnant women who received epidural analgesia in the first stage of labor,
* Pregnant women whose labor lasts less than 3 hours will not be included in the study.
* In case of any complications or cesarean section, the sample will be removed from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women will be included in the study.
Enrollment: 104 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Verbal Category Scale-VCS | pre-intervention
  VCS allows the person to describe pain by choosing the most appropriate expression. Using this scale, the pain experienced is categorized from mild to unbearable. They are numbered on the scale as Mild (1), Disturbing (2), Severe (3), Very Severe (4) and Unbearable (5). The patient is asked to choose the one that suits his/her condition from these options.
Visual Comparison Scale (VAS) | pre-intervention
  VAS is used to determine the patient's pain experience. A 10 cm long ruler is used for this purpose. At one end of this scale, there are "No Pain" categories and at the other end there are "Unbearable Pain" categories. It has been stated in the literature that this scale is more sensitive and reliable than other unidimensional scales. The patient is told that there are two end points and that he can mark any point he wishes among these points that is appropriate to the severity of his pain. The distance between the beginning of no pain and the point marked by the patient is measured and recorded in centimeters.
partograph | up to birth
  A partograph is a graphic record on paper that shows the progress of labor and indicates maternal and fetal status. It is helpful in recognizing cephalopelvic disproportion in labor that does not progress normally and in determining labor induction. It is an early warning system for labor induction, termination of labor, and the decision for caesarean section.
Evaluation of birth ball-VCS | immediately after the intervention
  VCS allows the person to describe pain by choosing the most appropriate expression. Using this scale, the pain experienced is categorized from mild to unbearable. They are numbered on the scale as Mild (1), Disturbing (2), Severe (3), Very Severe (4) and Unbearable (5). The patient is asked to choose the one that suits his/her condition from these options.
Evaluation of birth ball-satisfaction | up to 1-4 hours postpartum
  Mother Satisfaction Assessment Scale in Normal Birth: It was developed by Güngör and Beji and consists of 43 items and 10 subscales. Thirteen items (7,8,9,10,19,20,21,22,35,36,38,41,42) are reverse scored. The scale is a 5-point Likert type. It is scored as "1- I disagree, 2- I partially agree, 3- I am undecided, 4- I agree and 5- I strongly agree." As the total score from the scale increases, mothers' satisfaction level with the care they received in the hospital during normal birth increases.
Evaluation of birth dance-satisfaction | up to 1-4 hours postpartum
  Mother Satisfaction Assessment Scale in Normal Birth: It was developed by Güngör and Beji and consists of 43 items and 10 subscales. Thirteen items (7,8,9,10,19,20,21,22,35,36,38,41,42) are reverse scored. The scale is a 5-point Likert type. It is scored as "1- I disagree, 2- I partially agree, 3- I am undecided, 4- I agree and 5- I strongly agree." As the total score from the scale increases, mothers' satisfaction level with the care they received in the hospital during normal birth increases.
Evaluation of birth ball-VAS | immediately after the intervention
  Visual Comparison Scale (VAS): VAS is used to determine the patient's pain experience. A 10 cm long ruler is used for this purpose. At one end of this scale, there are "No Pain" categories and at the other end there are "Unbearable Pain" categories. It has been stated in the literature that this scale is more sensitive and reliable than other unidimensional scales. The patient is told that there are two end points and that he can mark any point he wishes among these points that is appropriate to the severity of his pain. The distance between the beginning of no pain and the point marked by the patient is measured and recorded in centimeters.
Evaluation of birth dance-VCS | immediately after the intervention
  VCS allows the person to describe pain by choosing the most appropriate expression. Using this scale, the pain experienced is categorized from mild to unbearable. They are numbered on the scale as Mild (1), Disturbing (2), Severe (3), Very Severe (4) and Unbearable (5). The patient is asked to choose the one that suits his/her condition from these options.
Evaluation of birth dance-VAS | immediately after the intervention
  Visual Comparison Scale (VAS): VAS is used to determine the patient's pain experience. A 10 cm long ruler is used for this purpose. At one end of this scale, there are "No Pain" categories and at the other end there are "Unbearable Pain" categories. It has been stated in the literature that this scale is more sensitive and reliable than other unidimensional scales. The patient is told that there are two end points and that he can mark any point he wishes among these points that is appropriate to the severity of his pain. The distance between the beginning of no pain and the point marked by the patient is measured and recorded in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Kılıç, Study Director — Ataturk University
Locations (1):
- Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital, Amasya, Center, Turkey (Türkiye)